CLINICAL TRIAL: NCT05358106
Title: A Phase 1, Single-blind, Partially Randomized, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Intravenous Doses of AntiBKV in Healthy Adult Volunteers.
Brief Title: Assess Safety, Tolerability and Pharmacokinetics of AntiBKV in Healthy Adult Volunteers.
Acronym: SAFE KIDNEY I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memo Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MTx-AntiBKV-AU-1.02BKVI
Record Dates: First submitted 2022-03-23; First posted 2022-05-03 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: BK Virus Nephropathy

STUDY DESIGN:
Intervention Model Description: Single-blind, partially randomized, placebo-controlled study in healthy volunteers. Approximately 40 to 56 healthy adult participants are planned to be enrolled in 7 cohorts of 4 to 8 participants, randomized in a 3:1 ratio to receive AntiBKV or placebo
Who Masked: Participant
Masking Description: Single-blind study where participants are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AntiBKV neutralising antibody (Active Comparator): AntiBKV infused i.v. over 30 minutes. Infusion parameters may be adjusted to bodyweight so that infusion rate does not exceed 60mg/kg per hour. AntiBKV will be administered as a single infusion in Part 1 or as 4 infusions administered 4 weeks apart in Part 2 (100, 500, 1000 or 2000 mg).
  Interventions: Biological: AntiBKV
- Placebo (Placebo Comparator): Solution containing no active excipients, infused i.v. over 30 minutes as a single infusion in Part 1 or as 4 infusions administered 4 weeks apart in Part 2.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AntiBKV — AntiBKV neutralising antibody
  Arms: AntiBKV neutralising antibody
Biological: Placebo — Solution with no active ingredients
  Arms: Placebo

SUMMARY:
BK virus (BKV) is a member of the polyomavirus family with a prevalence of up to 90% in the general population. In immunocompromized individuals, such as kidney transplant recipients (KTRs) who receive immunosuppressant therapy to prevent graft rejection, BKV turns into an opportunistic pathogen. BK viremia has been reported to occur in 10-30% of KTRs. BKV is recognized as a leading cause of impaired graft function and premature transplant loss, and is therefore a serious condition in kidney transplant patients.

At present, there are no effective agents specifically against BKV available and thus no standard treatment that can effectively reduce or prevent BKV infection/reactivation after renal transplantation. Therefore, the proposed indication for the AntiBKV neutralizing antibody is the treatment of BK virus infections and prevention of BK virus associated complications in KTRs.

This study has been designed to evaluate the safety, tolerability, and pharmacokinetic of ascending doses of AntiBKV, a fully human highly neutralising antibody against BKV, administered as a single or multiple intravenous infusions to healthy adult participants. The data obtained in this study will provide the basis for further clinical development of AntiBKV.

DETAILED DESCRIPTION:
BK virus (BKV) is a member of the polyomavirus family with a prevalence of up to 90% in the general population. It lies dormant and rarely causes disease in healthy individuals. However, in immunocompromized individuals, such as kidney transplant recipients (KTRs) who receive immunosuppressant therapy to prevent graft rejection, BKV turns into an opportunistic pathogen.

BKV replication can be detected before the development of BK virus associated nephropathy (BKVAN) and first virus shedding is detected in the urine. BK viremia has been reported to occur in 10-30% of KTRs. BKVAN progression is detected by a median of 8 weeks after establishment of the persistent viremia, and occurs most commonly in the first 2 years post-transplantation or following treatment of graft rejection. BKV infection/reactivation in these patients can lead to progression to BKVAN in up to 10% of all KTRs, while ultimately leading to graft dysfunction in 38% of patients and loss in 20% of patients presenting with BK viremia. BKV is recognized as a leading cause of impaired graft function and premature transplant loss, and is therefore a serious condition in kidney transplant patients.

At present, there are no effective agents specifically against BKV available and thus no standard treatment that can effectively reduce or prevent BKV infection/reactivation after renal transplantation.

The current standard of care after kidney transplantation involves prospective screening for BKV reactivation post-transplantation and subsequent reduction of immunosuppression to strengthen immune responses against BKV. Although reduction of immune suppression is a widely accepted management option, approaches for dose tapering differ with no consensus existing regarding when and which agent should be reduced or stopped following a diagnosis of BKV infection.

The proposed indication for the AntiBKV neutralizing antibody is the treatment of BK virus infections and prevention of BK virus associated complications in KTRs. In KTRs, the detection of the BK virus in the blood has been found to be strongly associated with the development of BKVAN and the grade of BK viremia correlates with the onset of the renal disease. A decrease of the virus load significantly reduces the chance for progression to BKVAN. Treatment of BK viremia with AntiBKV in KTRs with BKV infection/reactivation would allow for continued optimal immunosuppression to prevent graft rejection in these patients.

This study is the first clinical study to be conducted with AntiBKV and has been designed to evaluate the safety, tolerability, and pharmacokinetic of ascending doses of AntiBKV administered as single or multiple intravenous infusions to healthy adult participants. The data obtained in this study will provide the basis for further clinical development of AntiBKV.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged 18 years to 50 years at the time of consent
2. Ability to read, understand and provide written informed consent
3. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, including lifestyle restrictions for the duration of the study
4. Healthy participants as established by medical history, laboratory examination, physical examination, vital signs, and ECG during screening and as per the clinical judgment of the investigator
5. Body mass index (BMI) of 18.0 to 32.0 kg/m2 (inclusive)
6. For Woman of Childbearing Potential (WOCBP): agrees to practice true abstinence or agrees to use a highly effective method of contraception consistently from 30 days prior to Day 1 until at least 30 days post-dose. Highly effective contraception includes hormonal contraception, placement of intrauterine device (IUD) or intrauterine system (IUS), or a vasectomized partner (performed at least 6 months prior to her screening) who has been documented to no longer produce sperm. Verbal confirmation from the participant through medical interview is acceptable. No contraception requirements for participants in exclusive same-sex relationship.
7. For male participant: must agree to practice true abstinence or use condom if he has a partner of childbearing potential or must be surgically sterilized (performed at least 6 months prior and documented to no longer produce sperm. Verbal confirmation through medical interview is acceptable). Participant to practice abstinence (if applicable) or use condom for at least 30 days post-dose. No contraception requirements for participants in exclusive same-sex relationship.
8. Accessible veins in the forearms for venepuncture and/or intravenous cannulation

Exclusion Criteria:

1. Participant with active SARS-CoV-2 infection
2. Participants tested positive for human immunodeficiency virus (HIV antibody screen), Hepatitis B virus (HBsAg screen) or Hepatitis C virus (HCV antibody screen)
3. History of administration of any investigational or non-registered drug within 30 days or 5 half-lives, whichever is longer, prior to administration of study drug, or planned administration during the course of study participation.
4. History of any reaction to monoclonal antibodies.
5. History of allergic disease or reactions likely to be exacerbated by any component of the study drug, as assessed by the investigator, and/or known allergies to the trial product or its components.
6. History of any major pulmonary, cardiovascular, renal, neurological (e.g., cerebrovascular events), metabolic, gastrointestinal, hepato-biliary, or hematological functional abnormality, malignancy (except for adequately treated basal cell carcinoma or squamous cell carcinoma of the skin), or clinically significant mental disability that may interfere with the participant's ability to provide informed consent, as per discretion of the investigator. Gilbert's syndrome and history of cholecystectomy or cholecystitis will not be considered exclusionary.
7. Any abnormal laboratory finding at screening and at Day -1 (one retest is allowed at screening and/or at Day -1) unless deemed not clinically significant and irrelevant for study participation by the discretion of the investigator. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2 × upper limit of normal and/or glomerular filtration rate (GFR) <60ml/min are always considered exclusionary.
8. Acute illness (moderate or severe) and/or fever (body temperature ≥ 38 °C) during the 72 hours prior to any planned study drug application.
9. Participants with altered immunocompetence such as participants with ongoing cancer treatment, human immunodeficiency virus infection, organ transplant or any other active immune system disorder. Participants with seasonal allergies and mild asthma may be included.
10. Receipt of immunoglobulin or blood products within 6 months prior to enrolment.
11. Receipt of a monoclonal antibody within previous 6 months or 5 half-lives, whichever is longer.
12. Planned surgery (excluding minor procedures such as tooth extraction or incision and drainage) during the course of the study.
13. Receipt, or planned receipt of any standard vaccine within 7 days prior to and 7 days post Day 1 or planned vaccination within 7 days prior to and post any subsequent dosings.
14. History of alcoholism (>10 drinks/week) or drug addiction within 1 year prior to screening.
15. Positive screen for drugs of abuse or alcohol (breath test) at screening or Day -1 and prior to any subsequent dosings. A test may be repeated once at the discretion of the investigator to confirm suspected false-positive results.
16. Use of prescription drugs within 7 days prior to Day 1 or for 5 half-lives whichever is longer, or during the study, except for hormonal contraceptives.
17. Use of over-the-counter medication within 7 days prior to Day 1 or during the study; medication such as paracetamol and ibuprofen may be permitted at the discretion of the investigator and sponsor.
18. Receipt of immunosuppressive medications within 6 months prior to enrolment (receipt of any course of systemic corticosteroids for more than a 7-day duration and with a prednisolone equivalent dose of more than 5 mg per day within 6 months prior to enrolment will exclude a participant; inhaled or topical steroids are allowed).
19. Pregnant, lactating, or planned pregnancy during the study period.
20. Inability to comply with the study protocol in the opinion of the investigator.
21. Participant has any plans to permanently relocate from the area prior to the completion of the study or to leave for an extended period of time when study visits would need to be scheduled.
22. Concurrent participation in another interventional clinical study investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the study drug administration or during the course of the study.
23. Participant has clinically significant 12-lead ECG abnormalities at screening.
24. Abnormal vital signs including systolic blood pressure (SBP) < 90 or > 160 mmHg, diastolic blood pressure (DBP) < 50 or > 95 mmHg, heart rate (HR) < 45 or > 100 bpm (average of triplicate measurements) at screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To assess the number of participants with treatment related adverse events following a single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
Change in blood haematology values | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  Haematology data will be summarised for each scheduled visit, including observed values, change from baseline, number of out-of-range values and number of clinically significant values.
Change in blood biochemistry values | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  Biochemistry data will be summarised for each scheduled visit, including observed values, change from baseline, number of out-of-range values and number of clinically significant values.
Change in urinalysis values | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  Urinalysis data will be summarised for each scheduled visit, including observed values, change from baseline, number of out-of-range values and number of clinically significant values.
Change in blood pressure | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  Blood pressure results will be summarized for each scheduled timepoint, including observed values, change from baseline, number of out-of-range values and number of clinically significant values.
Change in heart rate | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  Heart rate will be summarized for each scheduled timepoint, including observed values, change from baseline, number of out-of-range values and number of clinically significant values.
Change in respiratory rate | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  Respiration rate will be summarized for each scheduled timepoint, including observed values, change from baseline, number of out-of-range values and number of clinically significant values.
Change in body temperature | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  Body temperature will be summarized for each scheduled timepoint, including observed values, change from baseline, number of out-of-range values and number of clinically significant values.
Participants with abnormal physical examination findings. | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  Abnormal physical examination findings during scheduled physical exams will be listed.
Change in P wave duration in electrocardiogram measurement | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  ECG parameters will be descriptively summarized for each scheduled timepoint, including observed values and change from baseline.
Change in PR interval in electrocardiogram measurement | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  ECG parameters will be descriptively summarized for each scheduled timepoint, including observed values and change from baseline.
Change in QRS duration in electrocardiogram measurement | Screening (Day -1) to final visit post-treatment (Day 113) for Part 1 and final visit post-treatment (Day 197) for Part 2.
  To evaluate the safety and tolerability of single ascending doses (Part 1) and multiple ascending doses (Part 2) of AntiBKV administered intravenously to healthy adult participants.
  ECG parameters will be descriptively summarized for each scheduled timepoint, including observed values and change from baseline.

SECONDARY OUTCOMES:
Pharmacokinetics measured by the maximum plasma concentration (Cmax) | Treatment Day 1 to final visit (Day 113) for Part 1 and final visit (Day 197) for Part 2.
  To assess the pharmacokinetic profile of AntiBKV in healthy participants after single (Part 1 and first dose in Part 2) or multiple (Part 2) intravenous dose administration.
Pharmacokinetics measured by the time of Cmax (Tmax) | Treatment Day 1 to final visit (Day 113) for Part 1 and final visit (Day 197) for Part 2.
  To assess the pharmacokinetic profile of AntiBKV in healthy participants after single (Part 1 and first dose in Part 2) or multiple (Part 2) intravenous dose administration.
Pharmacokinetics measured by the area under the curve (AUC) | Treatment Day 1 to final visit (Day 113) for Part 1 and final visit (Day 197) for Part 2.
  To assess the pharmacokinetic profile of AntiBKV in healthy participants after single (Part 1 and first dose in Part 2) or multiple (Part 2) intravenous dose administration.
Pharmacokinetics measured by the terminal elimination rate constant (λz) | Treatment Day 1 to final visit (Day 113) for Part 1 and final visit (Day 197) for Part 2.
  To assess the pharmacokinetic profile of AntiBKV in healthy participants after single (Part 1 and first dose in Part 2) or multiple (Part 2) intravenous dose administration.
Pharmacokinetics measured by the half life | Treatment Day 1 to final visit (Day 113) for Part 1 and final visit (Day 197) for Part 2.
  To assess the pharmacokinetic profile of AntiBKV in healthy participants after single (Part 1 and first dose in Part 2) or multiple (Part 2) intravenous dose administration.
Immunogenicity measured by anti-drug antibody (ADA) production | Treatment Day 1 to final visit (Day 113) for Part 1 and final visit (Day 197) for Part 2.
  Samples will be tested for the presence of ADAs. ADA titers and the presence of neutralizing antibodies will be determined for ADA positive samples

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Beck, Study Director — Memo Therapeutics AG
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
The Sponsor, MEMO Therapeutics AG., will not be sharing data with anyone outside of MEMO Therapeutics AG and the CRO involved in the study.

REFERENCES:
- [Derived] Helle F, Aubry A, Morel V, Descamps V, Demey B, Brochot E. Neutralizing Antibodies Targeting BK Polyomavirus: Clinical Importance and Therapeutic Potential for Kidney Transplant Recipients. J Am Soc Nephrol. 2024 Oct 1;35(10):1425-1433. doi: 10.1681/ASN.0000000000000457. Epub 2024 Jul 9. PMID 39352862